CLINICAL TRIAL: NCT02052193
Title: Evaluation of Photosensitivity in Dabrafenib or Vemurafenib Treated Metastatic Melanoma Patients - a Phase IIa/IIb Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Second cohort not opened because Simon-Two_Step model failed
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZDO 2012_PHOTOTOX
Record Dates: First submitted 2014-01-28; First posted 2014-01-31 (Estimated); Last update posted 2022-12-19 (Actual); Status verified 2015-07

CONDITIONS: Metastatic Melanoma (Carrying BRAF V600 Mutation)
MeSH Terms: conditions — Melanoma | interventions — dabrafenib; Vemurafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dabrafenib (Experimental): Dabrafenib 150mg BID orally
  Interventions: Drug: Dabrafenib; Drug: Vemurafenib
- Vemurafenib (Active Comparator): Vemurafenib 960mg orally BID
  Interventions: Drug: Dabrafenib; Drug: Vemurafenib

INTERVENTIONS:
Drug: Dabrafenib — Measurement of toxicity related to UV exposure
Drug: Vemurafenib — Measurement of toxicity related to UV exposure

SUMMARY:
The BRAF inhibitors dabrafenib and vemurafenib belong both two a new class of potent anti-cancer drugs and are highly efficacious in tumors harboring the BRAF V600E mutation. Both drugs seem to be equally efficacious; however, their toxicity profile seems to differ. Serious phototoxicity has been observed in ~ 30% of patients treated with vemurafenib and in ~2 percent of patients treated with dabrafenib. These phototoxic reactions have developed in spite of informing the patients of this possible adverse event and instructing them to protect themselves. Manifestation of phototoxic reactions depends on the patient's habits of exposure and their efforts to protect themselves. The true frequency of photosensitivity can only be established by systematic photo-testing. In dermatology, standard test procedures with different UV-wavelengths and dosages have been established and the primary goal of this study will be to clarify the true rate of photosensitivity by these two BRAF-inhibitors. Furthermore, systematic experience will be collected how to best protect patients from phototoxic events. Dabrafenib and Vemurafenib are commercially available and considered standard of care for BRAF mutant metastatic melanoma in Germany. As the number of patients will not allow any conclusion with regard to efficacy or safety of vemurafenib, patients randomized to vemurafenib in part 2 will only remain on study until completion of phototesting.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to performing any study-related procedures
* Male or female patients ≥ 18 years of age
* Patients with histologically confirmed metastatic melanoma (Stage III unresectable or Stage IV; American Joint Committee on Cancer, 7thEdition) with documented BRAF V600 mutation prior to first administration of dabrafenib or vemurafenib
* Patients must have measurable disease, defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 0.5 cm in the brain MRI with contrast
* ECOG performance status of 0 to 2
* Patients must have recovered from all side effects of their most recent systemic or local treatment for metastatic melanoma
* Adequate hematologic, renal, and liver function tests, as defined by the following laboratory values, performed within 7 days prior to first administration of dabrafenib or vemurafenib:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
  * Platelet count ≥ 100 x 109/L
  * Hemoglobin ≥ 9 g/dL
  * Serum creatinine ≤ 1.5 times upper limit of normal (ULN) or creatine clearance (CrCl) > 50 mL/min by Cockcroft-Gault formula
  * Aspartate aminotransferase (AST [SGOT]) and alanine aminotransferase (ALT [SGPT]) ≤ 2.5 times ULN
  * Serum bilirubin ≤ 1.5 times ULN
  * Alkaline phosphatase ≤ 2.5 times ULN (≤ 5 times ULN if considered due to liver metastases)
  * LVEF ≥ institutional LLN by ECHO
* Negative serum pregnancy test within 14 days prior to first administration of dabrafenib or vemurafenib in premenopausal women. Women of non-childbearing potential may be included if they are either surgically sterile or have been postmenopausal for ≥ 1 year
* Fertile women must use a highly effective method of contraception during treatment and for at least 1 month after completion of treatment, as directed by their physician. Effective methods of contraception are defined as those which result in a low failure rate (i.e., < 1% per year) when used consistently and correctly Hormonal-based methods (e.g., oral contraceptives) are not permitted due to potential drug-drug interactions with dabrafenib. See also "Pregnancy Testing and Prevention", page39. At the discretion of the investigator, acceptable methods of contraception may include total abstinence, in cases where the lifestyle of the patient ensures compliance. Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception
* Absence of any psychological, familial, sociological, or geographical conditions potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before trial entry
* Patients must be able to swallow tablets

Exclusion Criteria:

* Treatment with other UV sensitizing compounds such as psoralens, phenothiazine, tetracycline, amiodarone, phytopharmacons
* UV treatment within the last 3 months
* Previous treatment with a BRAF and/or MEK inhibitor.
* Cancer therapy (chemotherapy with delayed toxicity, extensive radiation therapy, immunotherapy, biologic therapy, or major surgery) within the last 3 weeks; chemotherapy regimens without delayed toxicity within the last 2 weeks; or use of an investigational anti-cancer drug within 28 days preceding the first dose of dabrafenib or vemurafenib
* Current use of a prohibited medication or requires any of these medications during treatment with dabrafenib or vemurafenib
* Current use of therapeutic warfarin NOTE: Low molecular weight heparin and prophylactic low-dose warfarin are permitted
* Unresolved toxicity of National Cancer Institute Common (NCI) Terminology Criteria for Adverse Events, v 4.0, ( Grade 2 or higher from previous anti-cancer therapy, except alopecia
* Presence of active gastrointestinal disease or other condition that will interfere significantly with the absorption of drugs
* A history of known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection
* Known immediate or delayed hypersensitivity reaction to Vemurafenib or Dabrafenib or excipients
* Presence of non-cutaneous malignancies other than metastatic melanoma (Stage IV) within 5 years of study enrollment or any malignancy with confirmed activating RAS mutation
* Brain metastases that are symptomatic and/or requiring corticosteroids. Subjects on a stable dose of corticosteroids >1 month or who have been off of corticosteroids for at least 2 weeks can be enrolled. Subjects must also be off of enzyme-inducing anticonvulsants for >4 weeks
* Corrected QT (QTc) interval >450 msecs; history of acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting within the past 24 weeks; Class II, III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system; abnormal cardiac valve morphology (≥ grade 2) documented by echocardiogram (subjects with minimal abnormalities [i.e., mild regurgitation/stenosis] can be entered on study with approval from the coordinating Investigator; or history of known cardiac arrhythmias
* Uncontrolled dysfunction of the electrolyte metabolism
* Known Long-QT-syndrome or intake of drugs which prolong the QT interval
* Uncontrolled medical conditions (i.e., diabetes mellitus, hypertension, etc.), psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol; or unwillingness or inability to follow the procedures required in the protocol
* Patients with extensive tattoos that would restrict skin surface available for phototesting or obscure skin reactions
* Pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12-15 (Actual)

PRIMARY OUTCOMES:
Degree of Solar Dermatitis due to Standardized UV Exposure in Patients treated with Dabrafenib | day 2-5
Degree of Solar Dermatitis due to Standardized UV Exposure in Patients treated with Dabrafenib or Vemurafenib | day 2-5

SECONDARY OUTCOMES:
Number of Participants with Adverse Events treated with dabrafenib | day 1-28
Best overall response rates and progression free survival in patients treated with dabrafenib or vemurafenib using RECIST v1.1 criteria | Every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Claus Garbe, M.D., Principal Investigator — Dept. of Dermatology, University Hopsital Tuebingen, Germany
Locations (1):
- Department of Dermatology, Tübingen, Baden-Wurttemberg, Germany